CLINICAL TRIAL: NCT00353730
Title: Identification of Genes Expressed in Atherosclerotic Plaques
Brief Title: Identification of Genes Expressed in Atherosclerotic Plaque
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020265; 02-H-0265
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis
Keywords: Serial Analysis of Gene Expression; Carotid Artery Plaque; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will identify genes and proteins in the blood of patients with atherosclerosis and in that of normal volunteers. The findings will be compared to determine the influence of these substances on the development of atherosclerosis a narrowing and hardening of blood vessel walls by deposits of fatty substances. Blood vessel blockage caused by atherosclerosis can impede blood flow and cause stroke, heart attack and poor limb circulation. The information from this study may lead to better ways to detect, prevent and treat these diseases.

Healthy volunteers and patients scheduled for carotid endarterectomy at Suburban Hospital in Bethesda, Maryland, are eligible for this study. Carotid endarterectomy is a surgical procedure in which the inner layer of the carotid artery (neck artery supplying blood to the brain) is scraped away to open the blocked vessel. Participants will undergo the following tests and procedures:

Patients

* Blood sample: Collection of about 32 cc (8 tablespoons) of blood for genetic and protein analysis
* Tissue sample: Collection of a piece of diseased blood vessel discarded from the endarterectomy procedure
* Review of records: Review of medical records for information about past illnesses, medications, tests, and so forth, if needed

Normal Volunteers

* Blood samples: Collection of about 32 cc (8 tablespoons) of blood for genetic and protein analysis
* Carotid artery ultrasound: Ultrasound imaging of the neck arteries for detection of any blockage
* Electrocardiogram: Recording of the electrical activity of the heart to detect any abnormalities in heart rhythm
* Echocardiogram: Ultrasound examination to detect possible abnormalities of the heart muscle
* Cardiac stress test: Treadmill stress test to detect possible heart vessel blockage (for subjects who have not had a cardiac stress test in the past year)
* Review of records: Review of medical records for information about past illnesses, medications, tests, and so forth, if needed

DETAILED DESCRIPTION:
Significant progress has been made in the prevention and treatment of atherosclerosis, but it continues to be a leading cause of morbidity and mortality in our society. The problem will become even more significant as an increasing proportion of the population ages. The goal of the proposed project is to advance our understanding of the genetic mechanisms of atherosclerosis. We propose to identify genes selectively expressed in peripheral monocytes of patients with atherosclerosis and in macrophages and endothelial cells of atherosclerotic plaques. We will examine gene expression profiles in purified subpopulations of cells using Serial Analysis of Gene Expression (SAGE) that requires only minute amounts of RNA, enabling the study of small homogeneous populations of cells. This sequence-based high-throughput gene expression profiling technique has the advantage of not requiring prior knowledge of the expressed gene sequences, allowing the discovery of new genes. With the completion of the human genome sequence, the SAGE technique is an ideal tool for comprehensively characterizing the transcriptomes of the important cells involved in atherosclerosis. This proposal is an exploratory study to find candidates, both known and unknown genes, which will be used for more extensive and statistically powered projects in the future. The insights obtained will be used for elucidating the pathogenesis of atherosclerosis and for developing new simple, sensitive and specific tests for early disease diagnosis. In addition, the new insights obtained may lead to the development of novel therapeutic strategies for disease prevention and treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any adult patient with carotid artery disease or known atherosclerosis capable of giving informed consent.

INCLUSION CRITERIA FOR MEDICATION TREATED SUBJECT:

Any adult with normal total cholesterol (less than 200 mg/dl) and blood pressure (systolic less than 140 and diastolic less than 90).

INCLUSION CRITERIA FOR NORMAL BRONCHOSCOPY SUBJECT:

Any healthy adult subject with no history of peripheral or coronary artery disease, who is eligible for bronchoalveolar lavage per Protocol 99-H-0068 and capable of giving informed consent.

EXCLUSION CRITERIA:

Unable to give consent

History of chronic infections, vasculitis or any other inflammatory disease

History of neoplastic disease or chemotherapy treatment

Immunosuppressive medications other than common over-the-counter drugs such as aspirin or acetaminophen

EXCLUSION CRITERIA FOR MEDICATION TREATED SUBJECT:

Subject with abnormal liver and renal function tests on pretreatment screening or currently taking a statin or ACE inhibitor medication.

EXCLUSION CRITERIA FOR NORMAL BRONCHOSCOPY SUBJECT:

Any exclusion criteria for normal subject listed in Protocol 99-H-0068.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2002-10-21 (Actual); Primary Completion 2005-03-16 (Actual); Study Completion 2011-01-12 (Actual)

PRIMARY OUTCOMES:
To identify known and unknown genes involved in the pathogenesis of atherosclerosis for further analyses. | ongoing
  To identify known and unknown genes involved in the pathogenesis of atherosclerosis.

SECONDARY OUTCOMES:
To identify atherosclerosis-specific genes expressed in peripheral monocytes, plaque macrophages or endothelial cells that may serve as early markers for disease diagnosis | ongoing
  To identify atherosclerosis-specific genes expressed in peripheral monocytes, plaque macrophages or endothelial cells that may serve as early markers for disease diagnosis
To identify genes expressed early in the pathogenesis of atherosclerosis that may be targeted for disease prevention. | ongoing
  To identify genes expressed early in the pathogenesis of atherosclerosis that may be targeted for disease prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Hwang, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Glass CK, Witztum JL. Atherosclerosis. the road ahead. Cell. 2001 Feb 23;104(4):503-16. doi: 10.1016/s0092-8674(01)00238-0. No abstract available. PMID 11239408
- [Background] Fayad ZA, Fuster V. Clinical imaging of the high-risk or vulnerable atherosclerotic plaque. Circ Res. 2001 Aug 17;89(4):305-16. doi: 10.1161/hh1601.095596. PMID 11509446
- [Background] Libby P, Ridker PM, Maseri A. Inflammation and atherosclerosis. Circulation. 2002 Mar 5;105(9):1135-43. doi: 10.1161/hc0902.104353. PMID 11877368
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-H-0265.html